CLINICAL TRIAL: NCT03787342
Title: Clinical and Radiographic Comparison of Double-Flap Incision, Modified Periosteal Releasing Incision, and Coronally Advanced Lingual Flap to Periosteal Releasing Incision for Flap Advancement in Partially Edentulous Patients Undergoing Guided Bone Regeneration Using Titanium Mesh: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Double-Flap Incision, Modified Periosteal Releasing Incision, and Coronally Advanced Lingual Flap to Periosteal Releasing Incision for Flap Advancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Zazou, Principle Investigator, assistant Lecturer, Modern Sciences and Arts University (MSA)., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERIO3:7:1
Record Dates: First submitted 2018-07-27; First posted 2018-12-26 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Flap Advancement
Keywords: Periosteal Releasing Incision, Modified Periosteal Releasing Incision, Coronally Advanced Lingual Flap, Double Flap Incision, Titanium mesh, GBR

STUDY DESIGN:
Intervention Model Description: Three Groups of intervention compared to one group of comparator. Each group contains 10 patients.
Who Masked: Participant, Outcomes Assessor
Masking Description: Care provider and investigator cannot be blinded as they are involved in the surgical procedure so blinding is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DFI "Double Flap Incision" (Experimental): A full-thickness crestal incision will be made over the edentulous ridge, and then one partial-thickness vertical incision will be made on the buccal side. A partial-thickness flap will be raised first to separate the mucosal layer from the overlying periosteum. Subsequently, the periosteal layer will be elevated to expose the underlying alveolar process. Xenograft and Ti-mesh will be used to augment the defective site then periosteal flap will be sutured first, with periosteal sutures securing the regenerative site. Then the mucosal flap will be closed.
  Interventions: Procedure: Double Flap Incision
- MPRI "Modified PRI" (Experimental): A full-thickness muco-periosteal flap is reflected on the buccal side (crestal incision and two vertical releasing incisions). Near the base of mucoperiosteal flap, the periosteum is incised less than 0.5mm in depth, creating two segments, "coronal segment" and "apical segment," of the periosteal flap. The shallow incision helps in preventing damage to the submucosal layer. The flap is pulled with a pair of periodontal forceps laterally. Subsequently, the "lateral stretching" of the coronal segment of the flap is performed by applying pressure using the blunt face of scalpel blade with sweeping motion to allow flap advancement.
  Interventions: Procedure: Modified Periosteal Releasing Incision
- CALF "Coronally Advanced Lingual Flap" (Experimental): A full-thickness crestal incision will be performed in the keratinized tissue from the distal surface of the more distal tooth to the retromolar pad. The flap design will be continued intrasulcularly on both vestibular and lingual sides of the mesial portion of the flap, buccally, it will be finished with a vertical releasing incision. On the lingual side, a full-thickness mucoperiosteal flap will be elevated until reaching the mylohyoid line. Then, using a blunt instrument it will be localized a connective tissue band continuing with the epimysium of the mylohyoid muscle. The blunt instrument will be inserted below this connective band, and, with gentle traction in the coronal direction, this muscular insertion will be detached from the lingual flap.
  Interventions: Procedure: Coronally Advanced Lingual Flap
- PRI "Periosteal Releasing Incision" (Active Comparator): A full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side and a full thickness flap will be raised. Xenograft and Ti-mesh will be used to augment the defective site then incremental incisions of 1-3 mm into the periosteum and submucosa will be used to advance the muco-periosteal flap. The flap will then be sutured as a whole unit.
  Interventions: Procedure: Periosteal releasing incision

INTERVENTIONS:
Procedure: Double Flap Incision — A full-thickness crestal incision will be made over the edentulous ridge, and then one partial-thickness vertical incision will be made on the buccal side. A partial-thickness flap will be raised first to separate the mucosal layer from the overlying periosteum. Subsequently, the periosteal layer will be elevated to expose the underlying alveolar process. Xenograft and Ti-mesh will be used to augment the defective site then periosteal flap will be sutured first, with periosteal sutures securing the regenerative site. Then the mucosal flap will be closed.
  Other Names: DFI
  Arms: DFI "Double Flap Incision"
Procedure: Modified Periosteal Releasing Incision — A full-thickness muco-periosteal flap is reflected on the buccal side (crestal incision and two vertical releasing incisions). Near the base of mucoperiosteal flap, the periosteum is incised less than 0.5mm in depth, creating two segments, "coronal segment" and "apical segment," of the periosteal flap. The shallow incision helps in preventing damage to the submucosal layer. The flap is pulled with a pair of periodontal forceps laterally. Subsequently, the "lateral stretching" of the coronal segment of the flap is performed by applying pressure using the blunt face of scalpel blade with sweeping motion to allow flap advancement.
  Other Names: MPRI
  Arms: MPRI "Modified PRI"
Procedure: Coronally Advanced Lingual Flap — A full-thickness crestal incision will be performed in the keratinized tissue from the distal surface of the more distal tooth to the retromolar pad. The flap design will be continued intrasulcularly on both vestibular and lingual sides of the mesial portion of the flap, buccally, it will be finished with a vertical releasing incision. On the lingual side, a full-thickness mucoperiosteal flap will be elevated until reaching the mylohyoid line. Then, using a blunt instrument it will be localized a connective tissue band continuing with the epimysium of the mylohyoid muscle. The blunt instrument will be inserted below this connective band, and, with gentle traction in the coronal direction, this muscular insertion will be detached from the lingual flap.
  Other Names: CALF
  Arms: CALF "Coronally Advanced Lingual Flap"
Procedure: Periosteal releasing incision
  Arms: PRI "Periosteal Releasing Incision"

SUMMARY:
Guided Bone Regeneration (GBR) is a reliable method to augment insufficient bone volume for implant placement. Membrane exposure is a major complication which is avoided by tension free primary closure. Classically Periosteal Releasing Incision (PRI) is performed to advance the flap. The aim of this trial is to compare Double Flap Incision (DFI), Modified Periosteal Releasing Incision (MPRI) & Coronally Advanced Lingual Flap (CALF) to PRI in terms of flap advancement, postoperative pain & swelling, membrane exposure and the amount of bone gain clinically and radiographically in GBR procedures.

DETAILED DESCRIPTION:
Study setting:

The patients will be assigned from the outpatient clinic of "The Faculty of Oral and Dental Medicine, Cairo University". Surgical procedures will be held in the periodontology clinic of the faculty. The recruited sample would be from the Egyptian urban and rural population.

Eligibility Criteria:

Inclusion criteria:

1. Partially edentulous patients in the mandibular posterior region.
2. Patients with healthy systemic condition.
3. Insufficient ridge width (< 5mm).
4. Presence of proper inter-arch space for placement of the implant prosthetic part.
5. Adequate soft tissue biotype (≥ 2mm).
6. No clinical evidence of active periodontal disease or oral infections.

Exclusion Criteria:

1. Patients with systemic conditions that may interfere with the results of the study.
2. Patients with local pathological defects related to the area of interest.
3. Unmotivated, uncooperative patients with poor oral hygiene.
4. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as smoking, alcoholism or para-functional habits.
5. History of bone associated diseases or medication affecting bone metabolism e.g.; bisphosphonate treatment.
6. History of radiation therapy in the head or neck region.
7. Current anti-tumor chemotherapy.
8. Pregnancy.
9. Inflammatory and autoimmune diseases of the oral cavity.

Interventions:

Pre-surgical phase:

1. Medical History Questionnaire (MHQ): Patients will be interviewed to gather information regarding general and oral health and MHQ will be filled by the patient and will be kept among patient's record file.
2. Clinical intra-oral examination

   * To ensure that the patient fulfills the previously mentioned defect-inclusion criteria.
   * Thorough intra-oral examination including teeth for caries, fracture, missing, or hopeless teeth and gingival-mucosal tissues for gingivitis, periodontitis, or oral lesions.
   * Referral for consultation or treatment if needed before the surgical phase.
3. If the patient meets the clinical selection criteria then radiographic examination will be held. CBCT will be performed for adequate evaluation of bone width and density and to be kept as a record for postoperative comparison.
4. Patients must sign an informed consent to clinical research previously approved by the Faculty of Oral and Dental Medicine, Cairo University.
5. Eligible patients will be randomized before being enrolled in the study.

Surgical phase:

The patients will be assigned into four groups, all undergoing GBR using Ti- mesh and Xenograft as follow:

* Group A: Flap advancement will be achieved using the DFI and this group will be assigned as a test group.
* Group B: Flap advancement will be achieved using the MPRI and this group will be assigned as a test group.
* Group C: Flap advancement will be achieved using the CALF and this group will be assigned as a test group.
* Group D: Flap advancement will be achieved using the PRI and this group will be assigned as the control group.

Surgical Protocol:

The surgical procedures will be performed under local anesthesia

Group A:

A full-thickness crestal incision will be made over the edentulous ridge, and then one partial-thickness vertical incision will be made on the buccal side. A partial-thickness flap will be raised first to separate the mucosal layer from the overlying periosteum. Subsequently, the periosteal layer will be elevated to expose the underlying alveolar process. Xenograft and Ti-mesh will be used to augment the defective site then periosteal flap will be sutured first, with periosteal sutures securing the regenerative site. Then the mucosal flap will be closed.

Group B:

A full-thickness muco-periosteal flap is reflected on the buccal side (crestal incision and two vertical releasing incisions). Near the base of mucoperiosteal flap, the periosteum is incised less than 0.5mm in depth, creating two segments, "coronal segment" and "apical segment," of the periosteal flap. The shallow incision helps in preventing damage to the submucosal layer. The flap is pulled with a pair of periodontal forceps laterally. Subsequently, the "lateral stretching" of the coronal segment of the flap is performed by applying pressure using the blunt face of scalpel blade with sweeping motion. This motion helps stretching the flap over the submucosa, thereby permitting the flap to be mobile and thus facilitates flap advancement (approximately 3-5mm). Xenograft and Ti-mesh will be used to augment the defective site.

Group C:

A full-thickness crestal incision will be performed in the keratinized tissue from the distal surface of the more distal tooth to the retromolar pad. The flap design will be continued intrasulcularly on both vestibular and lingual sides of the mesial portion of the flap, buccally, it will be finished with a vertical releasing incision. On the lingual side, a full-thickness mucoperiosteal flap will be elevated until reaching the mylohyoid line. Then, using a blunt instrument it will be localized a connective tissue band continuing with the epimysium of the mylohyoid muscle. The blunt instrument will be inserted below this connective band, and, with gentle traction in the coronal direction, this muscular insertion will be detached from the lingual flap.

Group D:

A full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side and a full thickness flap will be raised. Xenograft and Ti-mesh will be used to augment the defective site then incremental incisions of 1-3 mm into the periosteum and submucosa will be used to advance the muco-periosteal flap. The flap will then be sutured as a whole unit.

Post-surgical instructions:

* 1 g of Amoxicilin twice a day for 6 days with analgesic and anti-inflammatory drug, every 8 hours for 4 to 5 days, and 0.2% chlorexidine rinse 1min three times a day for 2 weeks, starting the day after surgery.
* Immediately after surgery, ice packs will be applied onto the treated area and it is recommended that they be kept in place for at least 4 h.
* Avoid tooth brushing especially at surgical sites, and soft diet to avoid trauma to the site of surgery for the first 3 weeks.
* Subsequent visits will be scheduled for healing assessment and measurement recording and if necessary, a professional supra-gingival prophylaxis will be performed.
* Sutures were removed after 2 week.
* A removable prosthesis was never allowed, during healing, to avoid trans-mucosal pressure on the operated area.

ELIGIBILITY:
Inclusion Criteria:

1. Partially edentulous patients in the mandibular posterior region.
2. Patients with healthy systemic condition.
3. Insufficient ridge width (< 5mm).
4. Presence of proper inter-arch space for placement of the implant prosthetic part.
5. Adequate soft tissue biotype (≥ 2mm).
6. No clinical evidence of active periodontal disease or oral infections.

Exclusion Criteria:

1. Patients with systemic conditions that may interfere with the results of the study.
2. Patients with local pathological defects related to the area of interest.
3. Unmotivated, uncooperative patients with poor oral hygiene.
4. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as smoking, alcoholism or para-functional habits.
5. History of bone associated diseases or medication affecting bone metabolism e.g.; bisphosphonate treatment.
6. History of radiation therapy in the head or neck region.
7. Current anti-tumor chemotherapy.
8. Pregnancy.
9. Inflammatory and autoimmune diseases of the oral cavity.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Flap advancement | Intraoperative
  Flap advancement in millimeters will be measured as the difference before and after Double flap Incision, Modified Periosteal Releasing Incision, Coronally Advanced Lingual Flap, and Periosteal Releasing Incision in millimeters using periodontal probe.

SECONDARY OUTCOMES:
Postoperative Pain | 7 days postoperatively
  Pain will be recorded using Numerical Rating scale (NRS). It is a scale from 0 to 10. 0 indicates no pain and 10 indicates severe pain.
Postoperative Swelling | 7 days postoperatively
  will be recorded using Visual Analogue Scale (VAS). It is a scale from 0 to 4. 0 indicates no swelling while 4 indicates severe extra-oral swelling.

OTHER OUTCOMES:
Postoperative membrane exposure | will be evaluated at 1, 2, 3, 4, 12, 24 weeks postoperative
  Measure the dimensions of the exposure using a periodontal probe in millimeters.
Bone width gain | preoperative & 6 months postoperative.
  The amount of bone gain will be measured before and after in millimeters on a cone beam CT & Clinically using bone caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Zazou, Masters, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt